CLINICAL TRIAL: NCT00110981
Title: A Multicenter, Open-Label, Pilot Trial to Evaluate the Effectiveness and Safety of ENBREL(r) in Combination With Narrowband UVB Phototherapy for the Treatment of Psoriasis
Brief Title: Utilization of Narrow Band Ultraviolet B (UVB) Light Therapy and Etanercept for the Treatment of Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040171
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Psoriasis
Keywords: psoriasis; dermatology; plaque psoriasis; skin; etanercept; ENBREL; NB-UVB, narrow-band UVB, phototherapy; combination therapy, 50 mg prefilled syringes
MeSH Terms: conditions — Psoriasis | interventions — Phototherapy; Etanercept

ARMS (1):
- Single-arm (Experimental)
  Interventions: Device: NB-UVB; Drug: Etanerept; Drug: Etanercept

INTERVENTIONS:
Device: NB-UVB — Three times a week (TIW) for 12 weeks
  Other Names: Phototherapy
Drug: Etanerept — 50 mg subcutaneously twice weekly (SC BIW) for 12 weeks
  Other Names: Enbrel
Drug: Etanercept — 50 mg subcutaneously twice weekly (SC BIW) for 12 weeks
  Other Names: Enbrel

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of combination therapy with etanercept and narrow-band (NB) UVB phototherapy for the treatment of psoriasis in a pilot study. This is a Phase 4 clinical study being conducted under an Amgen Investigational New Drug Application (IND).

ELIGIBILITY:
Inclusion Criteria: - Chronic plaque psoriasis eligible for systemic therapy and NB-UVB in the opinion of the investigator - Psoriasis Activity and Severity Index (PASI) greater than or equal to 15 and at least 25% of individual plaques must be considered severe - Patients must have body surface area (BSA) involvement of greater than or equal to 5% - Before any study-specific procedure, subject must sign and date the appropriate written informed consent - Negative urine pregnancy test within 7 days before the first dose of study drug in all women (except those surgically sterile or at least 5 years postmenopausal) - Sexually active subjects of childbearing potential must agree to use medically acceptable form of contraception during screening and throughout the study

Exclusion Criteria: - Prior phototherapy - Current or prior treatment with any tumor necrosis factor (TNF) antagonist, including etanercept, infliximab and adalimumab - Erythrodermic, pustular or guttate psoriasis - Evidence of skin conditions (e.g., eczema) other than psoriasis that would interfere with study-related evaluations of psoriasis - Evidence of active infections such as fevers, chills, sweats, or history of untreated Lyme disease and active severe infections within 4 weeks before screening visit or between the screening and baseline visits - History of immune compromised health [e.g., human immunodeficiency virus (HIV) positive status] - History of any cutaneous malignancy at any time, including squamous or basal cell carcinomas or melanoma - History of non-cutaneous cancer within 5 years - Actinic keratosis or atypical moles - History of alcohol or drug abuse within 12 months of screening visit - Current enrollment in another clinical study and treatment with another experimental drug or approved therapy for experimental use within 30 days prior to etanercept administration - Severe comorbidities as outlined in ENBREL(r) Package Insert: diabetes mellitus requiring insulin, congestive heart failure of any severity, myocardial infarction (within less than or equal to 52 weeks before screening), unstable angina pectoris, oxygen-dependent severe pulmonary disease, tuberculosis or tuberculosis exposure, chronic hepatitis B or hepatitis C, systemic lupus erythematosus, history of multiple sclerosis or other demyelinating disease, transverse myelitis, optic neuritis or epilepsy, uncontrolled hypertension (defined as systolic blood pressure greater than 180 mm Hg or diastolic blood pressure greater than 110 mm Hg) - Contraindications according to the ENBREL(r) Package Insert - Evidence of open cutaneous ulcers - Evidence of photosensitivity disorder (e.g., polymorphous light eruption) - Nursing mothers, female subjects planning on becoming pregnant or male subjects planning a pregnancy with their spouse/partner while in the study - Subjects that cannot commit to all the assessments required by the protocol - Known photosensitivity or known sensitivity to any of the excipients or products to be administered during dosing - Any disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-03; Primary Completion 2006-02 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving Psoriasis Area Severity Area (PASI) 75 at Week 12 | 3 months

SECONDARY OUTCOMES:
Time to PASI 75 responses | Variable
Proportion of subjects achieving PASI 90 at Week 12 | 3 months
Improvement in PASI at Week 12 | 3 months
Improvement in body surface area (BSA) involved with psoriasis at Week 12 | 3 months
Improvement in physician global assesssment of psoriasis, including an assessment of the proportion of subjects achieving clear or almost clear status at Week 12 | 3 months
Improvement in patient global assesssment of psoriasis at Week 12 | 3 months
Improvement in Dermatology Life Quality Index (DLQI) at Week 12 | 3 months
Subject incidence of serious adverse events (SAEs) and events of medical interests (EMI) at Week 12 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Kircik L, Bagel J, Korman N, Menter A, Elmets CA, Koo J, Yang YC, Chiou CF, Dann F, Stevens SR; Unite Study Group. Utilization of narrow-band ultraviolet light B therapy and etanercept for the treatment of psoriasis (UNITE): efficacy, safety, and patient-reported outcomes. J Drugs Dermatol. 2008 Mar;7(3):245-53. PMID 18380206
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20040171.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/